CLINICAL TRIAL: NCT03621670
Title: Safety and Immunogenicity of GSK Meningococcal Group B Vaccine and 13-valent Pneumococcal Vaccine Administered Concomitantly With Routine Infant Vaccines to Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205239; 2016-003268-37 (EudraCT Number); V72_57 (Other: Novartis)
Record Dates: First submitted 2018-07-10; First posted 2018-08-08 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Infections, Meningococcal
Keywords: Meningitis; Immune response; Sufficiency; Neisseria meningitides; Bexsero
MeSH Terms: conditions — Meningococcal Infections; Meningitis; Meningitis, Meningococcal | interventions — 4CMenB vaccine; PEDIARIX; Hiberix; RIX4414 vaccine; Measles-Mumps-Rubella Vaccine; Chickenpox Vaccine; Saline Waters

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind study Data are collected in an observer-blind manner. Observer-blind means that throughout the study, the participant/parent/caregiver, as well as site and sponsor personnel involved in the clinical evaluation of participants, are blinded, while other study personnel are aware of the treatment assignment. To maintain this blinding, authorized medical personnel prepare and administer the vaccines but do not participate in any clinical evaluation assays or procedures.
  Serological data that could lead to unblinding of the study groups are not available during the study to any investigator or personnel involved in the clinical conduct of the study. The laboratory responsible for the testing is blinded to the treatment, participant, and visit number, and uses coded identifiers to link the participant, visit, and study to each sample.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MenB+PCV Group (Experimental): Infant participants received rMenB+OMV NZ (Bexsero) along with PCV13 (Prevnar 13), Pediarix, Hiberix and Rotarix on Day 1 and Day 61 followed by rMenB+OMV NZ, PCV13, Pediarix and Hiberix on Day 121 and rMenB+OMV NZ, PCV13/PCV20, M-M-R II and Varivax on Day 301.
  Interventions: Biological: Bexsero (GSK Biologicals' Meningococcal group-B vaccine/ rMenB+OMV NZ); Biological: Prevnar13; Biological: Pediarix; Biological: Hiberix; Biological: Rotarix; Biological: M-M-R II; Biological: Varivax; Biological: Prevnar 20
- Placebo+PCV Group (Placebo Comparator): Infant participants received PCV13 along with placebo, Pediarix, Hiberix and Rotarix on Day 1 and Day 61 followed by PCV13, Placebo, Pediarix and Hiberix on Day 121 and PCV13/PCV20, Placebo M-M-R II and Varivax on Day 301.
  Interventions: Biological: Prevnar13; Biological: Pediarix; Biological: Hiberix; Biological: Rotarix; Biological: M-M-R II; Biological: Varivax; Biological: Placebo (saline water); Biological: Prevnar 20

INTERVENTIONS:
Biological: Bexsero (GSK Biologicals' Meningococcal group-B vaccine/ rMenB+OMV NZ) — Bexsero was administered intramuscularly on Day 1, Day 61, Day 121 and Day 301.
  Arms: MenB+PCV Group
Biological: Prevnar13 — Prevnar13 (PCV13) was administered intramuscularly on Day 1, Day 61, Day 121 and Day 301.
Biological: Pediarix — Pediarix (DTPa-HBV-IPV) was administered intramuscularly on Day 1, Day 61, and Day 121.
Biological: Hiberix — Hiberix (Hib) was administered intramuscularly on Day 1, Day 61, and Day 121.
Biological: Rotarix — Rotarix (HRV) was administered intramuscularly on Day 1 and Day 61.
Biological: M-M-R II — M-M-R II (MMR) was administered intramuscularly on Day 301.
Biological: Varivax — Varivax (VV) was administered intramuscularly on Day 301.
Biological: Placebo (saline water) — Placebo was administered intramuscularly on Day 1, Day 61, Day 121 and Day 301.
  Arms: Placebo+PCV Group
Biological: Prevnar 20 — Prevnar 20 (PCV13) was administered intramuscularly as a booster dose on Day 301 group who have received 3 PCV13 doses before 12 months of age but have not received their fourth booster dose.

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of Bexsero (meningococcal group B vaccine-rMenB+OMV NZ) in North American infants 6 weeks through 12 weeks of age, when administered concomitantly with Pneumococcal conjugate vaccine (PCV 13) and other recommended routine infant vaccinesv(RIV).

DETAILED DESCRIPTION:
This study is divided into three timepoints:

Epoch 1 - Primary: Day 1 to Day 301 Epoch 2 - Secondary: Day 301 to Day 331 Epoch 3 - Safety follow-up: Day 331 to the end of the study (Day 481 or Day 661). For participants who have not yet reached the 6-month safety follow-up after their last dose at the time Protocol Amendment 7 takes effect, visit 7 takes place on Day 481.

In addition to receiving the study vaccines, infants also receive non-study vaccines such as Diphtheria, tetanus toxoids and acellular pertussis adsorbed vaccine (DTPa, Infanrix) and Haemophilus influenzae type b Conjugate Vaccine (Hib, Hiberix) to minimize disruption to the standard infant vaccination schedule caused by participation in this study.

Participants receive rMenB+OMV NZ (Bexsero) concomitantly with PCV13 (Prevnar13) and other routine infant vaccines (Pediarix, Hiberix, Rotarix, M-M-R II, Varivax) at 2, 4, 6, and 12 months of age. Participants who have received three PCV13 doses before 12 months of age but have not yet received their fourth booster dose receive either PCV13 or PCV20 at 12 months of age (Visit 5).

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy all the following criteria at study entry:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol (e.g. completion of the eDiary, return for follow-up visits).
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to performing any study specific procedure.
* A male or female between, and including, 42 and 84 days of age (i.e., 6 through 12 weeks) at the time of the 1st vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born full-term (i.e. after a gestation period of ≥ 38 weeks).

Exclusion Criteria:

If any exclusion criterion applies, the subject must not be included in the study:

• Child in care

Each subject must not have:

* Progressive, unstable or uncontrolled clinical conditions.
* Hypersensitivity, including allergy to any component of vaccines, medicinal product or medical equipment whose use is foreseen in this study.
* Hypersensitivity to latex.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Abnormal function of the immune system resulting from:

  * Clinical conditions.
  * Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days from birth.
  * Administration of antineoplastic and immunomodulating agents or radiotherapy for any duration from birth.
  * Autoimmune disorders (including, but not limited to: blood, endocrine, hepatic, muscular, nervous system or skin autoimmune disorders; lupus erythematosus and associated conditions; rheumatoid arthritis and associated conditions; scleroderma and associated disorders) or immunodeficiency syndromes (including, but not limited to: acquired immunodeficiency syndromes and primary immunodeficiency syndromes).
* Received immunoglobulins or any blood products from birth.
* Received an investigational or non-registered medicinal product from birth.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.
* Neuroinflammatory disorders (including but not limited to: demyelinating disorders, encephalitis or myelitis of any origin), congenital and peripartum neurological conditions, encephalopathies, seizures (including all subtypes such as: absence seizures, generalised tonic-clonic seizures, partial complex seizures, partial simple seizures or febrile convulsions).
* Congenital or peripartum disorders resulting in a chronic condition (including but not limited to: chromosomal abnormalities, cerebral palsy, metabolism or synthesis disorders, cardiac disorders).
* Study personnel as an immediate family or household member.
* Current or previous, confirmed or suspected disease caused by N. meningitidis
* Household contact with and/or intimate exposure from birth to an individual with laboratory confirmed N. meningitidis and/or Streptococcus pneumoniae infection or colonization.
* Previous administration of meningococcal B or pneumococcal vaccine at any time prior to informed consent.
* Received a dose of DTPa-HBV-IPV, HRV, MMR, VV and/or Hib at any time prior to informed consent. Receipt of one dose of HBV up to 4 weeks prior to informed con-sent is allowed.
* Serious chronic illness.
* Uncorrected congenital malformation (such as Meckel's diverticulum) of the gastrointestinal tract that would predispose for Intussusception (IS).

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1196 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (51):
- United States (50):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Lake Mary, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Liverpool, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Boone, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Fairfield, Ohio
  - GSK Investigational Site, South Euclid, Ohio
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Edinburg, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Marshfield, Wisconsin
- GSK Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 1196 participants enrolled, only 1184 participants were included in the Exposed Set and started the study.
Period: Overall Study
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Started | 781 | 403
Completed | 642 | 326
Not Completed | 139 | 77
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 32 | 25
Not completed — Consent withdrawal not due to AEs | 54 | 18
Not completed — Migrated / Moved from the study area | 21 | 12
Not completed — Not willing / Not able to be contacted | 9 | 13
Not completed — Other | 13 | 5
Not completed — Protocol Deviation | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenB+PCV Group | Placebo+PCV Group | Total
Number analyzed (Participants) | 781 | 403 | 1184
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.6 (1.0) | 8.8 (1.0) | 8.7 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 380 | 196 | 576
  Male | 401 | 207 | 608
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17 | 4 | 21
  Asian | 39 | 21 | 60
  Black or African American | 84 | 33 | 117
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  White | 531 | 288 | 819
  Other (Not specified) | 107 | 56 | 163

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Events After the First Vaccination Administered at Day 1
Description: Assessed solicited administration site events include injection site tenderness (administration site pain), erythema (redness), swelling and induration. Any solicited administration site events = occurrence of the event regardless of intensity grade. Rotarix was administered orally; therefore, no administration site events were analyzed.
Time Frame: Day 1 to Day 7
Population: Analysis was performed on the Solicited Safety Set, which included all participants who received a study vaccination and had solicited adverse event data available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 768 | 394
Participants
  Erythema, Bexsero: number analyzed (Participants) | 768 | 0
  Erythema, Bexsero | 156 |
  Erythema, Prevnar 13: number analyzed (Participants) | 768 | 393
  Erythema, Prevnar 13 | 100 | 39
  Erythema, Placebo: number analyzed (Participants) | 0 | 394
  Erythema, Placebo |  | 25
  Erythema, Pediarix: number analyzed (Participants) | 768 | 391
  Erythema, Pediarix | 72 | 32
  Erythema, Hiberix: number analyzed (Participants) | 767 | 393
  Erythema, Hiberix | 74 | 17
  Induration, Bexsero: number analyzed (Participants) | 768 | 0
  Induration, Bexsero | 204 |
  Induration, Prevnar 13: number analyzed (Participants) | 768 | 393
  Induration, Prevnar 13 | 127 | 67
  Induration, Placebo: number analyzed (Participants) | 0 | 394
  Induration, Placebo |  | 22
  Induration, Pediarix: number analyzed (Participants) | 768 | 391
  Induration, Pediarix | 70 | 34
  Induration, Hiberix: number analyzed (Participants) | 767 | 393
  Induration, Hiberix | 77 | 20
  Swelling, Bexsero: number analyzed (Participants) | 768 | 0
  Swelling, Bexsero | 132 |
  Swelling, Prevnar 13: number analyzed (Participants) | 768 | 393
  Swelling, Prevnar 13 | 77 | 34
  Swelling, Placebo: number analyzed (Participants) | 0 | 394
  Swelling, Placebo |  | 21
  Swelling, Pediarix: number analyzed (Participants) | 768 | 391
  Swelling, Pediarix | 53 | 21
  Swelling, Hiberix: number analyzed (Participants) | 767 | 393
  Swelling, Hiberix | 54 | 12
  Tenderness, Bexsero: number analyzed (Participants) | 768 | 0
  Tenderness, Bexsero | 352 |
  Tenderness, Prevnar 13: number analyzed (Participants) | 768 | 393
  Tenderness, Prevnar 13 | 310 | 107
  Tenderness, Placebo: number analyzed (Participants) | 0 | 394
  Tenderness, Placebo | 0 | 81
  Tenderness, Pediarix: number analyzed (Participants) | 768 | 391
  Tenderness, Pediarix | 270 | 92
  Tenderness, Hiberix: number analyzed (Participants) | 767 | 393
  Tenderness, Hiberix | 284 | 74

2. Primary Outcome: Number of Participants Reporting Any Solicited Systemic Events After the First Vaccination Administered at Day 1
Description: Assessed systemic events include change in eating habits, sleepiness, vomiting, diarrhea, irritability, persistent crying, and fever, defined as body temperature greater than or equal to (≥)38.0°C/100.4°F. Any solicited systemic events = occurrence of the event regardless of intensity grade.
Time Frame: Day 1 to Day 7
Population: Analysis was performed on the Solicited Safety Set. Only participants with solicited adverse event data available for the specified duration were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 768 | 394
Participants
  Change in eating habits | 329 | 122
  Diarrhea | 173 | 84
  Irritability | 601 | 242
  Persistent crying | 248 | 89
  Sleepiness | 560 | 246
  Vomiting | 176 | 79
  Fever | 252 | 34

3. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Events After the Second Vaccination Administered at Day 61
Description: Rotarix was administered orally; therefore, no administration site events were analyzed.
Time Frame: Day 61 to Day 67
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 699 | 364
Participants
  Erythema, Bexsero: number analyzed (Participants) | 699 | 0
  Erythema, Bexsero | 200 |
  Erythema, Prevnar 13: number analyzed (Participants) | 697 | 363
  Erythema, Prevnar 13 | 129 | 62
  Erythema, Placebo: number analyzed (Participants) | 0 | 364
  Erythema, Placebo |  | 44
  Erythema, Pediarix: number analyzed (Participants) | 695 | 360
  Erythema, Pediarix | 99 | 54
  Erythema, Hiberix: number analyzed (Participants) | 697 | 363
  Erythema, Hiberix | 86 | 41
  Induration, Bexsero: number analyzed (Participants) | 699 | 0
  Induration, Bexsero | 213 |
  Induration, Prevnar 13: number analyzed (Participants) | 697 | 363
  Induration, Prevnar 13 | 142 | 63
  Induration, Placebo: number analyzed (Participants) | 0 | 364
  Induration, Placebo |  | 32
  Induration, Pediarix: number analyzed (Participants) | 695 | 360
  Induration, Pediarix | 109 | 55
  Induration, Hiberix: number analyzed (Participants) | 697 | 363
  Induration, Hiberix | 80 | 32
  Swelling, Bexsero: number analyzed (Participants) | 699 | 0
  Swelling, Bexsero | 112 |
  Swelling, Prevnar 13: number analyzed (Participants) | 697 | 363
  Swelling, Prevnar 13 | 74 | 38
  Swelling, Placebo: number analyzed (Participants) | 0 | 364
  Swelling, Placebo |  | 19
  Swelling, Pediarix: number analyzed (Participants) | 695 | 360
  Swelling, Pediarix | 52 | 33
  Tenderness, Bexsero: number analyzed (Participants) | 699 | 0
  Tenderness, Bexsero | 269 |
  Swelling, Hiberix: number analyzed (Participants) | 697 | 363
  Swelling, Hiberix | 49 | 17
  Tenderness, Prevnar 13: number analyzed (Participants) | 697 | 363
  Tenderness, Prevnar 13 | 227 | 81
  Tenderness, Placebo: number analyzed (Participants) | 0 | 364
  Tenderness, Placebo | 0 | 65
  Tenderness, Pediarix: number analyzed (Participants) | 695 | 360
  Tenderness, Pediarix | 201 | 67
  Tenderness, Hiberix: number analyzed (Participants) | 697 | 363
  Tenderness, Hiberix | 207 | 52

4. Primary Outcome: Number of Participants Reporting Any Solicited Systemic Events After the Second Vaccination Administered at Day 61
Time Frame: Day 61 to Day 67
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 699 | 364
Participants
  Change in eating habits | 238 | 90
  Diarrhea | 119 | 66
  Irritability | 514 | 215
  Persistent crying | 209 | 73
  Sleepiness | 455 | 183
  Vomiting | 104 | 49
  Fever | 269 | 64

5. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Events After the Third Vaccination Administered at Day 121
Time Frame: Day 121 to Day 127
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 676 | 352
Participants
  Erythema, Bexsero: number analyzed (Participants) | 676 | 0
  Erythema, Bexsero | 181 |
  Erythema, Prevnar 13: number analyzed (Participants) | 674 | 352
  Erythema, Prevnar 13 | 127 | 71
  Erythema, Placebo: number analyzed (Participants) | 0 | 351
  Erythema, Placebo |  | 43
  Erythema, Pediarix: number analyzed (Participants) | 672 | 351
  Erythema, Pediarix | 114 | 65
  Erythema, Hiberix: number analyzed (Participants) | 673 | 351
  Erythema, Hiberix | 97 | 38
  Induration, Bexsero: number analyzed (Participants) | 676 | 0
  Induration, Bexsero | 187 |
  Induration, Prevnar 13: number analyzed (Participants) | 674 | 352
  Induration, Prevnar 13 | 128 | 60
  Induration, Placebo: number analyzed (Participants) | 0 | 351
  Induration, Placebo |  | 26
  Induration, Pediarix: number analyzed (Participants) | 672 | 351
  Induration, Pediarix | 124 | 70
  Induration, Hiberix: number analyzed (Participants) | 673 | 351
  Induration, Hiberix | 86 | 28
  Swelling, Bexsero: number analyzed (Participants) | 676 | 0
  Swelling, Bexsero | 103 |
  Swelling, Prevnar 13: number analyzed (Participants) | 674 | 352
  Swelling, Prevnar 13 | 67 | 39
  Swelling, Placebo: number analyzed (Participants) | 0 | 351
  Swelling, Placebo |  | 13
  Swelling, Pediarix: number analyzed (Participants) | 672 | 351
  Swelling, Pediarix | 55 | 28
  Swelling, Hiberix: number analyzed (Participants) | 673 | 351
  Swelling, Hiberix | 36 | 8
  Tenderness, Bexsero: number analyzed (Participants) | 676 | 0
  Tenderness, Bexsero | 244 |
  Tenderness, Prevnar 13: number analyzed (Participants) | 674 | 352
  Tenderness, Prevnar 13 | 210 | 66
  Tenderness, Placebo: number analyzed (Participants) | 0 | 351
  Tenderness, Placebo |  | 52
  Tenderness, Pediarix: number analyzed (Participants) | 672 | 351
  Tenderness, Pediarix | 188 | 58
  Tenderness, Hiberix: number analyzed (Participants) | 673 | 351
  Tenderness, Hiberix | 194 | 45

6. Primary Outcome: Number of Participants Reporting Any Solicited Systemic Events After the Third Vaccination Administered at Day 121
Time Frame: Day 121 to Day 127
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 676 | 352
Participants
  Change in eating habits | 205 | 94
  Diarrhea | 87 | 44
  Irritability | 454 | 179
  Persistent crying | 151 | 59
  Sleepiness | 326 | 142
  Vomiting | 88 | 46
  Fever | 216 | 55

7. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Events After the Fourth Vaccination Administered at Day 301
Time Frame: Day 301 to Day 307
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 579 | 299
Participants
  Erythema, Bexsero: number analyzed (Participants) | 578 | 0
  Erythema, Bexsero | 180 |
  Erythema, Prevnar 13/20: number analyzed (Participants) | 564 | 288
  Erythema, Prevnar 13/20 | 119 | 37
  Erythema, Placebo: number analyzed (Participants) | 0 | 298
  Erythema, Placebo |  | 25
  Erythema, MMR II: number analyzed (Participants) | 569 | 294
  Erythema, MMR II | 64 | 24
  Erythema, Varivax: number analyzed (Participants) | 565 | 293
  Erythema, Varivax | 62 | 20
  Induration, Bexsero: number analyzed (Participants) | 579 | 0
  Induration, Bexsero | 179 |
  Induration, Prevnar 13/20: number analyzed (Participants) | 564 | 288
  Induration, Prevnar 13/20 | 109 | 32
  Induration, Placebo: number analyzed (Participants) | 0 | 298
  Induration, Placebo |  | 24
  Induration, MMR II: number analyzed (Participants) | 569 | 294
  Induration, MMR II | 46 | 17
  Induration, Varivax: number analyzed (Participants) | 565 | 293
  Induration, Varivax | 38 | 15
  Swelling, Bexsero: number analyzed (Participants) | 578 | 0
  Swelling, Bexsero | 91 |
  Swelling, Prevnar 13/20: number analyzed (Participants) | 564 | 287
  Swelling, Prevnar 13/20 | 52 | 18
  Swelling, Placebo: number analyzed (Participants) | 0 | 299
  Swelling, Placebo |  | 8
  Swelling, MMR II: number analyzed (Participants) | 569 | 294
  Swelling, MMR II | 26 | 12
  Swelling, Varivax: number analyzed (Participants) | 565 | 293
  Swelling, Varivax | 23 | 9
  Tenderness, Bexsero: number analyzed (Participants) | 579 | 0
  Tenderness, Bexsero | 223 |
  Tenderness, Prevnar 13/20: number analyzed (Participants) | 564 | 287
  Tenderness, Prevnar 13/20 | 181 | 35
  Tenderness, Placebo: number analyzed (Participants) | 0 | 298
  Tenderness, Placebo |  | 31
  Tenderness, MMR II: number analyzed (Participants) | 569 | 294
  Tenderness, MMR II | 130 | 28
  Tenderness, Varivax: number analyzed (Participants) | 565 | 293
  Tenderness, Varivax | 119 | 27

8. Primary Outcome: Number of Participants Reporting Any Solicited Systemic Events After the Fourth Vaccination Administered at Day 301
Time Frame: Day 301 to Day 307
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 614 | 314
Participants
  Change in eating habits: number analyzed (Participants) | 608 | 312
  Change in eating habits | 219 | 75
  Diarrhea: number analyzed (Participants) | 609 | 313
  Diarrhea | 85 | 40
  Irritability: number analyzed (Participants) | 614 | 313
  Irritability | 401 | 153
  Persistent crying: number analyzed (Participants) | 609 | 312
  Persistent crying | 115 | 29
  Rash: number analyzed (Participants) | 607 | 312
  Rash | 71 | 30
  Sleepiness: number analyzed (Participants) | 609 | 314
  Sleepiness | 273 | 96
  Vomiting: number analyzed (Participants) | 609 | 312
  Vomiting | 60 | 32
  Fever: number analyzed (Participants) | 608 | 312
  Fever | 118 | 22

9. Primary Outcome: Number of Participants With Any Solicited Systemic AEs During the 30 Days After the Fourth Vaccination at Day 301
Description: Systemic events assessed included rash, parotid/salivary gland swelling, and fever. These systemic adverse events were recorded for 30 days following MMR and VV vaccine administration. Any solicited systemic events = occurrence of the event regardless of intensity grade.
Time Frame: Day 301 to Day 330
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 627 | 321
Participants
  Parotid/Salivary gland swelling: number analyzed (Participants) | 626 | 321
  Parotid/Salivary gland swelling | 20 | 17
  Rash: number analyzed (Participants) | 626 | 321
  Rash | 206 | 95
  Fever | 197 | 70

10. Primary Outcome: Number of Participants Reporting Any Unsolicited Adverse Events (AEs) After the First Vaccination Administered at Day 1
Description: An unsolicited AEs is an AE that is not solicited using a subject diary and that is spontaneously communicated by the parent(s)/LAR(s) who has signed the informed consent or a solicited local or systemic AE that continues beyond the solicited period after vaccination. Any = occurrence of the event regardless of the intensity grade.
Time Frame: Day 1 to Day 30
Population: Analysis was performed on the Unsolicited Safety Set, which included all participants who received a study vaccination and had unsolicited adverse event data available for the specified duration
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 775 | 401
Participants | 214 | 103

11. Primary Outcome: Number of Participants Reporting Any Unsolicited AEs After the Second Vaccination Administered at Day 61
Time Frame: Day 61 to Day 90
Population: Analysis was performed on the Unsolicited Safety Set. Only participants with unsolicited adverse event data available for the specified duration were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 745 | 388
Participants | 225 | 119

12. Primary Outcome: Number of Participants Reporting Any Unsolicted AEs After the Third Vaccination Administered at Day 121
Time Frame: Day 121 to Day 150
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 725 | 374
Participants | 230 | 120

13. Primary Outcome: Number of Participants Reporting Any Unsolicited AEs After the Fourth Vaccination Administered at Day 301
Time Frame: Day 301 to Day 330
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 668 | 339
Participants | 248 | 144

14. Primary Outcome: Number of Participants Reporting Any SAEs, AEs Leading to Withdrawal, AESIs and MAAEs
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization and that results in disability/incapacity. An AE leading to withdrawal includes any AEs/SAEs collected and recorded from the time of the 1st receipt of study vaccines until study end which are identified as reasons for withdrawal of the participant from the study. AESIs are pre-defined (serious or non-serious) AEs of scientific and medical concern specific to the product or program which might warrant further investigation in order to characterize and understand it. MAAEs includes any AEs that required hospitalization, or an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits.
Time Frame: Day 1 up to study end (Day 481 for participants who have not reached 6-month follow-up at the time of Protocol Amendment 7; Day 661 for all others)
Population: Analysis was performed on the Unsolicited Safety Set. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 775 | 401
Participants
  AEs leading to withdrawal | 3 | 1
  SAEs | 35 | 19
  AESIs | 6 | 3
  MAAEs | 375 | 177

15. Primary Outcome: Percentage of Participants With Human Serum Bactericidal Assay (hSBA) Antibody Titers >= Lower Limit of Quantitation (LLOQ) for Each of the Serogroup B Test Strains M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4) and M13520 (NHBA)
Description: Serum bactericidal activity is assessed using human complement (hSBA) against Neisseria meningitidis serogroup B test strains: M14459 (fHbp); 96217 (NadA); NZ98/254 (PorA P1.4); M13520 (NHBA). The sufficiency of the immune response to rMenB+OMV NZ at one month after the third vaccination was to be demonstrated if the lower confidence limit for the percentage of participants achieving hSBA titers ≥ LLOQ is ≥ 60% for each of the M14459, 96217, NZ98/254, M13520 test strain. This outcome measure evaluated immune response to the rMenB+OMV NZ vaccine only, hence it was not applicable to the Placebo+PCV group.
Time Frame: At Day 151 (1 month after the third vaccination)
Population: Analysis was performed on the Per Protocol Set (PPS) for immunogenicity, which included all participants who received a study vaccination and provided immunogenicity data at one month after their third vaccination for at least 1 strain. Only participants with data available for the specified analysis at the specified timepoint were included.
Measure: Number (99.2% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 553
Percentage of participants
  M14459 (fHbp): number analyzed (Participants) | 537
  M14459 (fHbp) | 92.2 [88.6 to 94.9]
  96217 (NadA): number analyzed (Participants) | 525
  96217 (NadA) | 99.4 [97.9 to 99.9]
  NZ98/254 (PorA): number analyzed (Participants) | 547
  NZ98/254 (PorA) | 73.5 [68.2 to 78.3]
  M13520 (NHBA) | 53.0 [47.3 to 58.6]

16. Primary Outcome: Percentage of Participants With hSBA Titers >= LLOQ Against All Serogroup B Test Strains Combined (Composite Response)
Description: The immune response to the rMenB+OMV NZ vaccine is assessed by measuring serum bactericidal activity using hSBA against four Neisseria meningitidis serogroup B test strains: M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA). The composite response is defined as the percentage of participants with hSBA titers ≥ Lower Limit of Quantitation (LLOQ) across all four strains combined. The sufficiency of the immune response to rMenB+OMV NZ at one month after the third vaccination was to be demonstrated if the lower confidence limit for the percentage of participants achieving hSBA titers ≥ LLOQ is ≥ 50% for all strains combined. This outcome measure evaluated immune response to the rMenB+OMV NZ vaccine only, hence it was not applicable to the Placebo+PCV group.
Time Frame: At Day 151 (1 month after the third vaccination)
Population: Analysis was performed on the PPS for immunogenicity. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Number (99.2% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 524
Percentage of participants | 42.7 [37.0 to 48.6]

17. Primary Outcome: Percentage of Participants With hSBA Antibody Titers >= 8 for Strains M14459 (fHbp); 96217 (NadA); NZ98/254 (PorA P1.4); M13520 (NHBA) and >= 16 for Strain 96217
Description: Serum bactericidal activity is assessed using human complement (hSBA) against Neisseria meningitidis serogroup B test strains: M14459 (fHbp); 96217 (NadA); NZ98/254 (PorA P1.4); M13520 (NHBA). The sufficiency of the immune response to rMenB+OMV NZ at one month after the 4th vaccination was to be demonstrated if the lower confidence limit for the percentage of participants achieving hSBA titers ≥ 8 (for strains M14459, NZ98/254, M13520) and ≥16 (for strain 96217) is ≥75% for each of the M14459, 96217, NZ98/254, M13520 test strains. This outcome measure evaluated immune response to the rMenB+OMV NZ vaccine only, hence it was not applicable to the Placebo+PCV group.
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Number (95.8% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 505
Percentage of participants
  M14459 (fHbp): number analyzed (Participants) | 492
  M14459 (fHbp) | 89.0 [85.8 to 91.7]
  96217 (NadA): number analyzed (Participants) | 482
  96217 (NadA) | 99.6 [98.5 to 100]
  NZ98/254 (PorA P1.4): number analyzed (Participants) | 499
  NZ98/254 (PorA P1.4) | 83.2 [79.4 to 86.5]
  M13520 (NHBA) | 76.6 [72.5 to 80.4]

18. Primary Outcome: Percentage of Participants With hSBA Antibody Titers >= 8 for Strains M14459 (fHbp), NZ98/254 (PorA P1.4), and M13520 (NHBA) and >= 16 for Strain 96217 (NadA) (Composite Response Across All Strains)
Description: The immune response to the rMenB+OMV NZ vaccine is assessed by measuring serum bactericidal activity using hSBA against four Neisseria meningitidis serogroup B test strains: M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA). The composite response is defined as the percentage of participants with hSBA titers ≥ Lower Limit of Quantitation (LLOQ) across all four strains combined. The sufficiency of the immune response to rMenB+OMV NZ at one month after the 4th vaccination was to be demonstrated if the lower confidence limit for the percentage of participants achieving hSBA titers ≥ 8 (for strains M14459, NZ98/254, M13520) and ≥16 (for strain 96217) is ≥65% for all strains combined. This outcome measure evaluated immune response to the rMenB+OMV NZ vaccine only, hence it was not applicable to the Placebo+PCV group.
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Number (95.8% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 478
Percentage of participants | 63.2 [58.5 to 67.7]

19. Primary Outcome: Adjusted Geometric Mean Concentrations (GMCs) of Immunoglobubin (IgG) Antibodies Against 13 PCV13 Antigens at 1 Month After Third Vaccination
Description: The immune response to PCV13 is evaluated by measuring IgG levels using electrochemiluminescence (ECL) assay. Adjusted GMCs are assessed for each of the 13 PCV13 antigens at 1 month after the third vaccination.
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Geometric Mean (98.3% Confidence Interval); unit: Microgram per milliliter(µg/mL)
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 244 | 278
Microgram per milliliter(µg/mL)
  Serotype 1 | 1.6 [1.4 to 1.9] | 1.5 [1.3 to 1.8]
  Serotype 3 | 0.5 [0.4 to 0.6] | 0.5 [0.4 to 0.6]
  Serotype 4 | 1.1 [0.9 to 1.3] | 1.1 [1.0 to 1.3]
  Serotype 5 | 1.0 [0.8 to 1.2] | 1.0 [0.8 to 1.2]
  Serotype 6 | 2.4 [2.0 to 2.8] | 2.5 [2.1 to 2.9]
  Serotype 6B | 1.5 [1.1 to 1.9] | 1.8 [1.4 to 2.3]
  Serotype 7F | 2.8 [2.4 to 3.3] | 2.9 [2.5 to 3.3]
  Serotype 9V | 1.3 [1.1 to 1.6] | 1.4 [1.2 to 1.6]
  Serotype 14 | 5.9 [4.7 to 7.4] | 5.8 [4.8 to 7.2]
  Serotype 18C | 1.5 [1.3 to 1.8] | 1.5 [1.3 to 1.8]
  Serotype 19A | 1.7 [1.4 to 2.0] | 1.8 [1.6 to 2.2]
  Serotype 19F | 2.5 [2.1 to 2.9] | 2.5 [2.2 to 2.9]
  Serotype 23F: number analyzed (Participants) | 244 | 277
  Serotype 23F | 0.9 [0.7 to 1.1] | 1.0 [0.8 to 1.2]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of PCV13 when administered concomitantly with rMenB+OMV NZ and other RIV, compared to PCV13 and other RIV alone without rMenB+OMV NZ, at one month after the third vaccination; Test type: Non-Inferiority — The non-inferiority (NI) was to be demonstrated if the lower limit of the 2-sided 98.3% confidence interval (CI) of the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 1 antigen; Group GMC Ratio = 1.05, 98.3% CI 2-sided [0.90 to 1.23] — GMCs and alpha-adjusted CIs were derived by exponentiating (base 10) the least squares means and 95% CI of log10-transformed antibody concentrations from a two-way Analysis of Variance (ANOVA), accounting for vaccine-group and center effects
Statistical Analysis 2: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 3 antigen; Group GMC Ratio = 0.90, 98.3% CI 2-sided [0.77 to 1.06] — GMCs and alpha-adjusted CIs were derived by exponentiating (base 10) the least squares means and 95% CI of log10-transformed antibody concentrations from a two-way ANOVA, accounting for vaccine-group and center effects
Statistical Analysis 3: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 4 antigen; Group GMC Ratio = 0.98, 98.3% CI 2-sided [0.84 to 1.15] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 4: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 5 antigen; Group GMC Ratio = 1.03, 98.3% CI 2-sided [0.86 to 1.22] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 5: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 6 antigen; Group GMC Ratio = 0.95, 98.3% CI 2-sided [0.81 to 1.11] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 6: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 6B antigen; Group GMC Ratio = 0.80, 98.3% CI 2-sided [0.63 to 1.02] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 7: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 7F antigen; Group GMC Ratio = 0.98, 98.3% CI 2-sided [0.85 to 1.12] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 8: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 9V antigen; Group GMC Ratio = 0.94, 98.3% CI 2-sided [0.80 to 1.12] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 9: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 14 antigen; Group GMC Ratio = 1.01, 98.3% CI 2-sided [0.82 to 1.24] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 10: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 18C antigen; Group GMC Ratio = 1.00, 98.3% CI 2-sided [0.85 to 1.18] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 11: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 19A antigen; Group GMC Ratio = 0.91, 98.3% CI 2-sided [0.77 to 1.06] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 12: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 19F antigen; Group GMC Ratio = 0.99, 98.3% CI 2-sided [0.86 to 1.14] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 13: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 19, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 98.3% CI for the between-group ratio of ECL assay GMC is >0.5 for the PCV13 Serotype 23F antigen; Group GMC Ratio = 0.87, 98.3% CI 2-sided [0.73 to 1.05] — [estimate comment as in outcome 19, analysis 2]

20. Secondary Outcome: Adjusted GMCs of IgG Antibodies Against 13 PCV13 Antigens at 1 Month After the Fourth Vaccination Administered at Day 301
Description: The immune response to PCV13 is evaluated by measuring IgG levels using ECL assay. Adjusted GMCs are assessed for each of the 13 PCV13 antigens at 1 month after the 4th vaccination.
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 225 | 240
µg/mL
  Serotype 1 | 1.8 [1.5 to 2.1] | 1.8 [1.6 to 2.1]
  Serotype 3: number analyzed (Participants) | 225 | 239
  Serotype 3 | 0.5 [0.4 to 0.6] | 0.5 [0.5 to 0.6]
  Serotype 4 | 1.5 [1.2 to 1.8] | 1.7 [1.4 to 2.0]
  Serotype 5 | 1.8 [1.5 to 2.1] | 1.8 [1.6 to 2.1]
  Serotype 6 | 5.2 [4.4 to 6.1] | 6.0 [5.2 to 7.0]
  Serotype 6B | 4.7 [3.9 to 5.6] | 5.4 [4.6 to 6.4]
  Serotype 7F | 3.7 [3.2 to 4.4] | 4.6 [4.0 to 5.3]
  Serotype 9V: number analyzed (Participants) | 224 | 240
  Serotype 9V | 2.3 [2.0 to 2.8] | 2.6 [2.2 to 3.1]
  Serotype 14 | 7.0 [5.8 to 8.4] | 7.1 [6.0 to 8.4]
  Serotype 18C | 2.0 [1.7 to 2.4] | 2.2 [1.9 to 2.6]
  Serotype 19A | 4.5 [3.8 to 5.3] | 5.5 [4.7 to 6.4]
  Serotype 19F | 4.8 [4.1 to 5.7] | 5.0 [4.3 to 5.9]
  Serotype 23F | 1.9 [1.5 to 2.3] | 1.9 [1.6 to 2.3]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of PCV13 when administered concomitantly with rMenB+OMV NZ and other RIV, compared to PCV13 and other RIV alone, at one month after the fourth vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 1 antigen; Group GMC Ratio = 0.95, 95% CI 2-sided [0.82 to 1.11] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 2: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 3 antigen; Group GMC Ratio = 0.90, 95% CI 2-sided [0.79 to 1.03] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 3: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 4 antigen; Group GMC Ratio = 0.90, 95% CI 2-sided [0.77 to 1.07] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 4: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 5 antigen; Group GMC Ratio = 0.97, 95% CI 2-sided [0.83 to 1.12] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 5: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 6 antigen; Group GMC Ratio = 0.86, 95% CI 2-sided [0.74 to 0.99] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 6: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 6B antigen; Group GMC Ratio = 0.86, 95% CI 2-sided [0.73 to 1.02] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 7: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 7F antigen; Group GMC Ratio = 0.81, 95% CI 2-sided [0.70 to 0.93] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 8: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 9V antigen; Group GMC Ratio = 0.90, 95% CI 2-sided [0.77 to 1.06] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 9: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 14 antigen; Group GMC Ratio = 0.99, 95% CI 2-sided [0.83 to 1.17] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 10: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 18C antigen; Group GMC Ratio = 0.89, 95% CI 2-sided [0.76 to 1.04] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 11: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 19A antigen; Group GMC Ratio = 0.82, 95% CI 2-sided [0.71 to 0.95] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 12: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 19F antigen; Group GMC Ratio = 0.96, 95% CI 2-sided [0.83 to 1.12] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 13: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group ratio of ECL assay GMCs is >0.5 for the PCV13 Serotype 23F antigen; Group GMC Ratio = 0.97, 95% CI 2-sided [0.82 to 1.16] — [estimate comment as in outcome 19, analysis 2]

21. Secondary Outcome: Percentage of Participants With Serum Pneumococcal Anti-capsular Polysaccharide IgG >= 0.35 μg/mL
Description: The immune response to PCV13 is evaluated by measuring the percentage of participants with serum IgG concentrations ≥ 0.35 μg/mL for each of the 13 PCV13 antigens at 1 month after the third and fourth vaccinations.
Time Frame: At Day 151 (1 month after the third vaccination) and Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 244 | 278
Percentage of participants
  Serotype 1, At Day 151 | 99.2 [97.1 to 99.9] | 97.1 [94.4 to 98.7]
  Serotype 1, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 1, At Day 331 | 98.7 [96.2 to 99.7] | 97.1 [94.1 to 98.8]
  Serotype 3, At Day 151 | 59.8 [53.4 to 66.0] | 61.5 [55.5 to 67.3]
  Serotype 3, At Day 331: number analyzed (Participants) | 225 | 239
  Serotype 3, At Day 331 | 63.6 [56.9 to 69.8] | 69.5 [63.2 to 75.2]
  Serotype 4, At Day 151 | 94.3 [90.6 to 96.8] | 96.0 [93.0 to 98.0]
  Serotype 4, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 4, At Day 331 | 97.8 [94.9 to 99.3] | 96.7 [93.5 to 98.6]
  Serotype 5, At Day 151 | 91.0 [86.7 to 94.3] | 87.4 [82.9 to 91.1]
  Serotype 5, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 5, At Day 331 | 96.0 [92.5 to 98.2] | 98.8 [96.4 to 99.7]
  Serotype 6, At Day 151 | 99.2 [97.1 to 99.9] | 99.6 [98.0 to 100]
  Serotype 6, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 6, At Day 331 | 100 [98.4 to 100] | 99.6 [97.7 to 100]
  Serotype 6B, At Day 151 | 89.8 [85.2 to 93.3] | 92.4 [88.7 to 95.3]
  Serotype 6B, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 6B, At Day 331 | 100 [98.4 to 100] | 99.6 [97.7 to 100]
  Serotype 7F, At Day 151 | 99.6 [97.7 to 100] | 100 [98.7 to 100]
  Serotype 7F, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 7F, At Day 331 | 99.6 [97.5 to 100] | 100 [98.5 to 100]
  Serotype 9V, At Day 151 | 95.1 [91.6 to 97.4] | 93.2 [89.5 to 95.8]
  Serotype 9V, At Day 331: number analyzed (Participants) | 224 | 240
  Serotype 9V, At Day 331 | 98.7 [96.1 to 99.7] | 98.8 [96.4 to 99.7]
  Serotype 14, At Day 151 | 98.0 [95.3 to 99.3] | 98.6 [96.4 to 99.6]
  Serotype 14, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 14, At Day 331 | 100 [98.4 to 100] | 100 [98.5 to 100]
  Serotype 18C, At Day 151 | 97.5 [94.7 to 99.1] | 96.8 [93.9 to 98.5]
  Serotype 18C, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 18C, At Day 331 | 99.1 [96.8 to 99.9] | 99.2 [97.0 to 99.9]
  Serotype 19A, At Day 151 | 96.7 [93.6 to 98.6] | 98.6 [96.4 to 99.6]
  Serotype 19A, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 19A, At Day 331 | 100 [98.4 to 100] | 99.6 [97.7 to 100]
  Serotype 19F, At Day 151 | 99.6 [97.7 to 100] | 100 [98.7 to 100]
  Serotype 19F, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 19F, At Day 331 | 100 [98.4 to 100] | 100 [98.5 to 100]
  Serotype 23F, At Day 151: number analyzed (Participants) | 244 | 277
  Serotype 23F, At Day 151 | 87.3 [82.5 to 91.2] | 87.0 [82.5 to 90.7]
  Serotype 23F, At Day 331: number analyzed (Participants) | 225 | 240
  Serotype 23F, At Day 331 | 97.3 [94.3 to 99.0] | 97.1 [94.1 to 98.8]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of PCV13 when administered concomitantly with rMenB+OMV NZ and other RIV, compared to PCV13 and other RIV alone, at one month after the third vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 1 antigen; Difference in percentage = 2.06, 95% CI 2-sided [-0.38 to 4.87] — The 95% CI of the between MenB+PCV and Placebo+PCV group-difference has been derived using the method of Miettinen and Nurminen
Statistical Analysis 2: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 1]; Difference in percentage = 1.58, 95% CI 2-sided [-1.28 to 4.74] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 3 antigen; Difference in percentage = -1.67, 95% CI 2-sided [-10.07 to 6.70] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 20, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 3]; Difference in percentage = -5.90, 95% CI 2-sided [-14.45 to 2.69] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 5: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of PCV13 when administered concomitantly with rMenB+OMV NZ and other RIV compared to PCV13 and other RIV alone, at one month after the third vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 4 antigen; Difference in percentage = -1.78, 95% CI 2-sided [-5.87 to 1.97] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 6: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of PCV13 when administered concomitantly with rMenB+OMV NZ and other RIV compared to PCV13 and other RIV alone, at one month after the fourth vaccination; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 5]; Difference in percentage = 1.11, 95% CI 2-sided [-2.17 to 4.51] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 7: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 5 antigen; Difference in percentage = 3.57, 95% CI 2-sided [-1.86 to 8.96] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 8: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 7]; Difference in percentage = -2.75, 95% CI 2-sided [-6.33 to 0.16] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 9: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 6 antigen; Difference in percentage = -0.46, 95% CI 2-sided [-2.62 to 1.27] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 10: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 9]; Difference in percentage = 0.42, 95% CI 2-sided [-1.27 to 2.33] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 11: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 6B antigen; Difference in percentage = -2.69, 95% CI 2-sided [-7.86 to 2.21] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 12: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 11]; Difference in percentage = 0.42, 95% CI 2-sided [-1.27 to 2.33] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 13: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 7F antigen; Difference in percentage = -0.41, 95% CI 2-sided [-2.29 to 0.96] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 14: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 13]; Difference in percentage = -0.44, 95% CI 2-sided [-2.48 to 1.14] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 15: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 9V antigen; Difference in percentage = 1.92, 95% CI 2-sided [-2.30 to 6.12] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 16: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 15]; Difference in percentage = -0.09, 95% CI 2-sided [-2.76 to 2.44] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 17: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 14 antigen; Difference in percentage = -0.61, 95% CI 2-sided [-3.43 to 1.87] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 18: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 17]; Difference in percentage = 0.00, 95% CI 2-sided [-1.68 to 1.58] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 19: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 18C antigen; Difference in percentage = 0.78, 95% CI 2-sided [-2.40 to 3.91] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 20: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 19]; Difference in percentage = -0.06, 95% CI 2-sided [-2.44 to 2.20] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 21: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 19A antigen; Difference in percentage = -1.84, 95% CI 2-sided [-5.06 to 0.83] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 22: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 21]; Difference in percentage = 0.42, 95% CI 2-sided [-1.27 to 2.33] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 23: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 19F antigen; Difference in percentage = -0.41, 95% CI 2-sided [-2.29 to 0.96] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 24: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 23]; Difference in percentage = 0.00, 95% CI 2-sided [-1.68 to 1.58] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 25: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 5]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with IgG ≥ 0.35 µg/mL is >-10% for the PCV13 Serotype 23F antigen; Difference in percentage = 0.29, 95% CI 2-sided [-5.62 to 6.07] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 26: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 21, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 21, analysis 25]; Difference in percentage = 0.25, 95% CI 2-sided [-3.13 to 3.58] — [estimate comment as in outcome 21, analysis 1]

22. Secondary Outcome: Adjusted GMCs Against 3 Pertussis Antigens (Pertussis Toxin [PT], Pertactin [PRN], Filamentous Hemagglutinin [FHA])
Description: The immune response to DTaP-HBV-IPV (Pediarix) vaccine is evaluated. IgG concentrations for pertussis antigens (PT, FHA, PRN) are measured at 1 month after the third vaccination and are expressed as international units per millilitre (IU/mL).
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 470 | 266
IU/mL
  PT: number analyzed (Participants) | 468 | 266
  PT | 50.3 [45.1 to 56.0] | 59.6 [53.2 to 66.8]
  FHA | 106.7 [96.4 to 118.0] | 133.1 [119.5 to 148.2]
  Pertactin | 41.7 [36.1 to 48.1] | 65.7 [56.4 to 76.4]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of DTaP-HBV-IPV vaccine when administered concomitantly with rMenB+OMV NZ and PCV13 compared to DTaP-HBV-IPV vaccine concomitantly administered with PCV13 without rMenB+OMV NZ, in terms of PT, FHA and PRN, at one month after the third vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group GMC ratio is >0.67 for the antigen PT; Group GMC Ratio = 0.84, 95% CI 2-sided [0.76 to 0.94] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 2: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 22, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group GMC ratio is >0.67 for the antigen FHA; Group GMC Ratio = 0.80, 95% CI 2-sided [0.73 to 0.88] — [estimate comment as in outcome 19, analysis 2]
Statistical Analysis 3: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 22, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group GMC ratio is >0.67 for the antigen PRN; Group GMC Ratio = 0.63, 95% CI 2-sided [0.55 to 0.73] — [estimate comment as in outcome 19, analysis 2]

23. Secondary Outcome: Percentage of Participants With Antibodies Concentrations Against Hepatitis B Surface Antigen (AntiHBsAg) >= 10 mIU/mL
Description: The immune response to DTaP-HBV-IPV vaccine administered with rMenB+OMV NZ and PCV13 is evaluated. IgG concentrations for Hepatitis B (HepB) antigens are measured at 1 month after the third vaccination.
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 105 | 138
Percentage of participants | 100 [96.5 to 100] | 99.3 [96.0 to 100]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of DTaP-HBV-IPV vaccine when administered concomitantly with rMenB+OMV NZ and PCV13 compared to DTaP-HBV-IPV vaccine concomitantly administered with PCV13 without rMenB+OMV NZ, in terms of Hep B, at one month after the third vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with anti-HBs >=10 mIU/mL is >-10% for the HBs antigen; Difference in percentage = 0.72, 95% CI 2-sided [-2.83 to 4.00] — [estimate comment as in outcome 21, analysis 1]

24. Secondary Outcome: Percentage of Participants With Anti-diphtheria and Anti-tetanus Antibody Concentrations >= 0.1 IU/mL
Description: The immune response to DTaP-HBV-IPV vaccine administered with rMenB+OMV NZ and PCV13 is evaluated. IgG concentrations for diphtheria (D) and tetanus (T) were measured at 1 month after the third vaccination.
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 224 | 143
Percentage of participants
  Tetanus Toxoid | 100 [98.4 to 100] | 100 [97.5 to 100]
  Diphtheria Toxoid: number analyzed (Participants) | 220 | 136
  Diphtheria Toxoid | 99.5 [97.5 to 100] | 100 [97.3 to 100]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of DTaP-HBV-IPV vaccine when administered concomitantly with rMenB+OMV NZ and PCV13 compared to DTaP-HBV-IPV vaccine concomitantly administered with PCV13 without rMenB+OMV NZ, in terms of D, at one month after the third vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with anti-diphtheria toxoid concentrations >=0.1 IU/mL is >-10%; Difference in percentage = 0.00, 95% CI 2-sided [-1.69 to 2.62] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of DTaP-HBV-IPV vaccine when administered concomitantly with rMenB+OMV NZ and PCV13 compared to DTaP-HBV-IPV vaccine concomitantly administered with PCV13 without rMenB+OMV NZ, in terms of T, at one month after the third vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with anti-tetanus toxoid concentrations >=0.1 IU/mL is >-5%; Difference in percentage = -0.45, 95% CI 2-sided [-2.53 to 2.30] — [estimate comment as in outcome 21, analysis 1]

25. Secondary Outcome: Percentage of Participants With Anti-polyribosyl-ribitol Phosphate (PRP) Concentration >= 0.15 µg/mL and >= 1 µg/mL
Description: The immune response to Hib vaccine administered with rMenB+OMV NZ and PCV13 is evaluated. IgG concentrations for Haemophilus influenzae type b (Hib) are measured at 1 month after the third vaccination.
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 347 | 264
Percentage of participants
  >= 0.15 µg/mL | 98.3 [96.3 to 99.4] | 97.7 [95.1 to 99.2]
  >= 1 µg/mL | 87.0 [83.0 to 90.4] | 84.1 [79.1 to 88.3]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of Hib vaccine when administered concomitantly with rMenB+OMV NZ and PCV13 compared to Hib vaccine concomitantly administered with PCV13 without rMenB+OMV NZ, in terms of Hib, at one month after the third vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with anti-PRP concentration >=0.15 µg/mL is >-5%; Difference in percentage = 0.54, 95% CI 2-sided [-1.79 to 3.32] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 25, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the group differences in percentage of participants with anti-PRP concentration >=1 µg/mL is >-10%; Difference in percentage = 2.94, 95% CI 2-sided [-2.63 to 8.78] — [estimate comment as in outcome 21, analysis 1]

26. Secondary Outcome: Adjusted GMCs for Anti-measles Antibodies
Description: The immune response to MMR vaccine administered with rMenB+OMV NZ and PCV13 is evaluated. IgG concentrations for measles antigens are measured using adjusted GMCs at 1 month after fourth vaccination and are expressed as milli-International Units per milliliter (mIU/mL).
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 435 | 235
mIU/mL | 877.3 [743.7 to 1035.0] | 873.5 [732.2 to 1042.0]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of MMR vaccine when administered concomitantly with rMenB+OMV NZ and PCV13 compared to MMR vaccine concomitantly administered with PCV13, without rMenB+OMV NZ, at one month after fourth vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group GMC ratio is > 0.67 for the antigen "Measles"; Group GMC Ratio = 1.00, 95% CI 2-sided [0.86 to 1.17] — [estimate comment as in outcome 19, analysis 2]

27. Secondary Outcome: Adjusted GMCs for Anti-mumps Antibodies
Description: The immune response to MMR vaccine administered with rMenB+OMV NZ and PCV13 is evaluated. IgG concentrations for mumps antigens are measured using adjusted GMCs at 1 month after fourth vaccination.
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units per milliliter (AU/mL)
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 435 | 235
Arbitrary Units per milliliter (AU/mL) | 744.5 [628.5 to 882.0] | 856.8 [715.0 to 1026.7]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; [analysis description as in outcome 26, analysis 1]; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group GMC ratio is > 0.67 for the antigen "Mumps"; Group GMC Ratio = 0.87, 95% CI 2-sided [0.74 to 1.02] — [estimate comment as in outcome 19, analysis 2]

28. Secondary Outcome: Adjusted GMCs for Anti-rubella Antibodies
Description: The immune response to MMR vaccine administered with rMenB+OMV NZ and PCV13 is evaluated. IgG concentrations for rubella antigens are measured using adjusted GMCs at 1 month after fourth vaccination.
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 432 | 235
IU/mL | 57.7 [50.0 to 66.6] | 54.0 [46.3 to 63.0]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of MMR vaccine when administered concomitantly with rMenB+OMV NZ, VV and PCV13 compared to MMR vaccine concomitantly administered with PCV13, without rMenB+OMV NZ, at one month after fourth vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group GMC ratio is > 0.67 for the antigen "Rubella"; Group GMC Ratio = 1.07, 95% CI 2-sided [0.93 to 1.22] — [estimate comment as in outcome 19, analysis 2]

29. Secondary Outcome: Adjusted GMCs for Anti-Varicella (VV) Antibodies
Description: The immune response to varicella (VV) vaccine administered with rMenB+OMV NZ and PCV13 is evaluated. IgG concentrations for varicella antigens are measured using GMCs at 1 month after fourth vaccination.
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 437 | 231
mIU/mL | 1283.8 [1137.4 to 1449.2] | 1208.9 [1060.5 to 1378.2]
Statistical Analysis 1: Comparison: MenB+PCV Group vs Placebo+PCV Group; To demonstrate the immunological non-inferiority of VV vaccine when administered concomitantly with rMenB+OMV NZ, MMR and PCV13 compared to VV vaccine concomitantly administered with PCV13, without rMenB+OMV NZ, at one month after fourth vaccination; Test type: Non-Inferiority — The NI was to be demonstrated if the lower limit of the 2-sided 95% CI for the between-group GMC ratio is > 0.67 for the antigen "VZV gE"; Group GMC Ratio = 1.06, 95% CI 2-sided [0.95 to 1.19] — [estimate comment as in outcome 19, analysis 2]

30. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >= 5, >= 8 and >=16 for Each of the Serogroup B Test Strains M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA)
Description: This immune response to the rMenB+OMV NZ vaccine only is evaluated, hence it was not applicable to the Placebo+PCV group.
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 553
Percentage of participants
  M14459 (fHbp), >= 5: number analyzed (Participants) | 537
  M14459 (fHbp), >= 5 | 92.2 [89.6 to 94.3]
  M14459 (fHbp), >= 8: number analyzed (Participants) | 537
  M14459 (fHbp), >= 8 | 82.9 [79.4 to 86.0]
  M14459 (fHbp), >= 16: number analyzed (Participants) | 537
  M14459 (fHbp), >= 16 | 50.5 [46.2 to 54.8]
  96217 (NadA), >= 5: number analyzed (Participants) | 525
  96217 (NadA), >= 5 | 99.6 [98.6 to 100]
  96217 (NadA), >= 8: number analyzed (Participants) | 525
  96217 (NadA), >= 8 | 99.6 [98.6 to 100]
  96217 (NadA), >= 16: number analyzed (Participants) | 525
  96217 (NadA), >= 16 | 99.4 [98.3 to 99.9]
  NZ98/254 (PorA P1.4), >= 5: number analyzed (Participants) | 547
  NZ98/254 (PorA P1.4), >= 5 | 77.7 [74.0 to 81.1]
  NZ98/254 (PorA P1.4), >= 8: number analyzed (Participants) | 547
  NZ98/254 (PorA P1.4), >= 8 | 61.8 [57.6 to 65.9]
  NZ98/254 (PorA P1.4), >= 16: number analyzed (Participants) | 547
  NZ98/254 (PorA P1.4), >= 16 | 31.1 [27.2 to 35.1]
  M13520 (NHBA), >= 5 | 60.4 [56.2 to 64.5]
  M13520 (NHBA), >= 8 | 32.4 [28.5 to 36.4]
  M13520 (NHBA), >= 16 | 9.4 [7.1 to 12.1]

31. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >= 5 and >= 8 for Each of the Serogroup B Test Strains M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA)
Description: as for outcome 30
Time Frame: At Day 301 (6 months after third vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 540
Percentage of participants
  M14459 (fHbp), >= 5: number analyzed (Participants) | 516
  M14459 (fHbp), >= 5 | 14.5 [11.6 to 17.9]
  M14459 (fHbp), >= 8: number analyzed (Participants) | 516
  M14459 (fHbp), >= 8 | 4.8 [3.2 to 7.1]
  96217 (NadA) >= 5: number analyzed (Participants) | 505
  96217 (NadA) >= 5 | 97.8 [96.1 to 98.9]
  96217 (NadA), >= 8: number analyzed (Participants) | 505
  96217 (NadA), >= 8 | 96.4 [94.4 to 97.9]
  NZ98/254 (PorA P1.4), >= 5: number analyzed (Participants) | 531
  NZ98/254 (PorA P1.4), >= 5 | 20.2 [16.8 to 23.8]
  NZ98/254 (PorA P1.4), >= 8: number analyzed (Participants) | 531
  NZ98/254 (PorA P1.4), >= 8 | 12.2 [9.6 to 15.3]
  M13520 (NHBA), >= 5 | 10.2 [7.8 to 13.1]
  M13520 (NHBA) >= 8 | 5.9 [4.1 to 8.3]

32. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >= 5 for Each of the Serogroup B Test Strain M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA)
Description: as for outcome 30
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 505
Percentage of participants
  M14459 (fHbp), >= 5: number analyzed (Participants) | 492
  M14459 (fHbp), >= 5 | 94.5 [92.1 to 96.4]
  96217 (NadA), >= 5: number analyzed (Participants) | 482
  96217 (NadA), >= 5 | 99.6 [98.5 to 99.9]
  NZ98/254 (PorA P1.4), >= 5: number analyzed (Participants) | 499
  NZ98/254 (PorA P1.4), >= 5 | 89.6 [86.6 to 92.1]
  M13520 (NHBA), >= 5 | 91.5 [88.7 to 93.8]

33. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against Each of the Serogroup B Test Strains M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA)
Description: as for outcome 30
Time Frame: At Day 151 (1 month after the third vaccination), Day 301 (6 months after the third vaccination), and Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 553
Titer
  M14459 (fHbp), Day 151: number analyzed (Participants) | 537
  M14459 (fHbp), Day 151 | 15.1 [13.7 to 16.7]
  M14459 (fHbp), Day 301: number analyzed (Participants) | 516
  M14459 (fHbp), Day 301 | 3.0 [2.8 to 3.2]
  M14459 (fHbp), Day 331: number analyzed (Participants) | 492
  M14459 (fHbp), Day 331 | 24.3 [21.3 to 27.8]
  96217 (NadA), Day 151: number analyzed (Participants) | 525
  96217 (NadA), Day 151 | 488.2 [437.3 to 545.0]
  96217 (NadA), Day 301: number analyzed (Participants) | 505
  96217 (NadA), Day 301 | 89.1 [77.3 to 102.7]
  96217 (NadA), Day 331: number analyzed (Participants) | 482
  96217 (NadA), Day 331 | 1349.0 [1195.3 to 1522.5]
  NZ98/254 (PorA P1.4), Day 151: number analyzed (Participants) | 547
  NZ98/254 (PorA P1.4), Day 151 | 10.1 [8.9 to 11.4]
  NZ98/254 (PorA P1.4), Day 301: number analyzed (Participants) | 531
  NZ98/254 (PorA P1.4), Day 301 | 3.8 [3.5 to 4.0]
  NZ98/254 (PorA P1.4), Day 331: number analyzed (Participants) | 499
  NZ98/254 (PorA P1.4), Day 331 | 20.3 [17.3 to 23.7]
  M13520 (NHBA), Day 151 | 5.5 [5.0 to 6.0]
  M13520 (NHBA), Day 301: number analyzed (Participants) | 540
  M13520 (NHBA), Day 301 | 3.5 [3.3 to 3.7]
  M13520 (NHBA), Day 331: number analyzed (Participants) | 505
  M13520 (NHBA), Day 331 | 12.7 [11.2 to 14.4]

34. Secondary Outcome: hSBA Geometric Mean Ratios (GMRs) Over Pre Fourth Vaccination Against Each of the Serogroup B Test Strains M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA)
Description: as for outcome 30
Time Frame: At Day 331 (1 month after the fourth vaccination) compared to Day 301 (pre-fourth vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 465
Ratio
  M14459 (fHbp): number analyzed (Participants) | 435
  M14459 (fHbp) | 8.7 [7.6 to 10.0]
  96217 (NadA): number analyzed (Participants) | 420
  96217 (NadA) | 17.4 [15.1 to 20.1]
  NZ98/254 (PorA P1.4): number analyzed (Participants) | 452
  NZ98/254 (PorA P1.4) | 5.5 [4.7 to 6.5]
  M13520 (NHBA) | 3.9 [3.4 to 4.4]

35. Secondary Outcome: Percentage of Participants With hSBA Antibody Titers >= LLOQ for Each of the Serogroup B Test Strains M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA)
Description: as for outcome 30
Time Frame: At Day 301 (6 months after the third vaccination) and Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 540
Percentage of participants
  M14459 (fHbp), Day 301: number analyzed (Participants) | 516
  M14459 (fHbp), Day 301 | 14.5 [11.6 to 17.9]
  M14459 (fHbp), Day 331: number analyzed (Participants) | 492
  M14459 (fHbp), Day 331 | 94.5 [92.1 to 96.4]
  96217 (NadA), Day 301: number analyzed (Participants) | 505
  96217 (NadA), Day 301 | 94.1 [91.6 to 96.0]
  96217 (NadA), Day 331: number analyzed (Participants) | 482
  96217 (NadA), Day 331 | 99.6 [98.5 to 99.9]
  M13520 (NHBA), Day 301 | 8.5 [6.3 to 11.2]
  M13520 (NHBA), Day 331: number analyzed (Participants) | 505
  M13520 (NHBA), Day 331 | 86.1 [82.8 to 89.0]
  NZ98/254 (PorA P1.4), Day 301: number analyzed (Participants) | 531
  NZ98/254 (PorA P1.4), Day 301 | 17.5 [14.4 to 21.0]
  NZ98/254 (PorA P1.4), Day 331: number analyzed (Participants) | 499
  NZ98/254 (PorA P1.4), Day 331 | 87.6 [84.4 to 90.3]

36. Secondary Outcome: Percentage of Participants With 4-fold Rise in hSBA Titers for Each of the Serogroup B Test Strains M14459 (fHbp), 96217 (NadA), NZ98/254 (PorA P1.4), and M13520 (NHBA)
Description: A 4-fold rise in hSBA titers is defined as - if pre-vaccination titer <Limit of Detection (LOD), then a post-vaccination titer >= 4 times the LOD or >= LLOQ, whichever is greater; - if pre-vaccination titer is >= LOD but <LLOQ, then a post-vaccination titer >= 4 times the LLOQ; - if pre-vaccination titer is >= LLOQ, then a post-vaccination titer >= 4 times the pre-vaccination titer, where pre-vaccination titer=pre-4th dose titers (Day 301). This outcome measure evaluated immune response to the rMenB+OMV NZ vaccine only, hence it was not applicable to the Placebo+PCV group.
Time Frame: At Day 331 (1 month after the fourth vaccination) relative to Day 301 (pre-fourth vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group
Number analyzed (Participants) | 465
Percentage of participants
  M14459 (fHbp), Day 331: number analyzed (Participants) | 435
  M14459 (fHbp), Day 331 | 72.0 [67.5 to 76.1]
  96217 (NadA), Day 331: number analyzed (Participants) | 420
  96217 (NadA), Day 331 | 94.8 [92.2 to 96.7]
  M13520 (NHBA), Day 331 | 36.1 [31.8 to 40.7]
  NZ98/254 (PorA P1.4), Day 331: number analyzed (Participants) | 452
  NZ98/254 (PorA P1.4), Day 331 | 54.2 [49.5 to 58.9]

37. Secondary Outcome: Percentage of Participants With Anti-HBs Antibody Concentrations >= 100 mIU/mL
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 105 | 138
Percentage of participants | 98.1 [93.3 to 99.8] | 96.4 [91.7 to 98.8]

38. Secondary Outcome: GMCs for Anti-HBsAg Antibodies
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 105 | 138
mIU/mL | 2201.0 [1554.7 to 3116.0] | 2404.8 [1803.1 to 3207.3]

39. Secondary Outcome: Percentage of Participants With Anti-diphtheria and Anti-tetanus Antibody Concentrations >= 1 IU/mL
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 224 | 143
Percentage of participants
  Tetanus Toxoid | 67.0 [60.4 to 73.1] | 69.2 [61.0 to 76.7]
  Diphtheria Toxoid: number analyzed (Participants) | 220 | 136
  Diphtheria Toxoid | 40.0 [33.5 to 46.8] | 55.1 [46.4 to 63.7]

40. Secondary Outcome: GMCs for Anti-diphtheria and Anti-tetanus Antibodies
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 224 | 143
IU/mL
  Tetanus Toxoid | 1.5 [1.3 to 1.8] | 1.6 [1.3 to 1.9]
  Diphtheria Toxoid: number analyzed (Participants) | 220 | 136
  Diphtheria Toxoid | 0.9 [0.8 to 1.1] | 1.2 [1.0 to 1.5]

41. Secondary Outcome: Percentage of Participants With Anti-polio Type 1, 2 and 3 Neutralization Antibody Titers >= 8
Time Frame: At Day 151 (1 month after the third vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 106 | 120
Percentage of participants
  Polio 1: number analyzed (Participants) | 102 | 120
  Polio 1 | 100 [96.4 to 100] | 100 [97.0 to 100]
  Polio 2: number analyzed (Participants) | 106 | 116
  Polio 2 | 99.1 [94.9 to 100] | 100 [96.9 to 100]
  Polio 3: number analyzed (Participants) | 97 | 112
  Polio 3 | 100 [96.3 to 100] | 99.1 [95.1 to 100]

42. Secondary Outcome: Percentage of Participants With Seroresponse for Anti-Varicella (VV), Anti-measles Virus, Anti-mumps Virus and Anti-rubella Virus Antibodies
Description: Seroresponse is defined as post-vaccination anti-VZV virus, anti-measles virus, anti-mumps virus and anti-rubella virus antibody concentration >= a protective threshold among participants who were seronegative (antibody concentration < assay cut-off) before vaccination.
Time Frame: At Day 331 (1 month after the fourth vaccination)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MenB+PCV Group | Placebo+PCV Group
Number analyzed (Participants) | 364 | 201
Percentage of participants
  Mumps: number analyzed (Participants) | 354 | 198
  Mumps | 81.6 [77.2 to 85.5] | 85.9 [80.2 to 90.4]
  Measles: number analyzed (Participants) | 347 | 191
  Measles | 94.8 [91.9 to 96.9] | 97.9 [94.7 to 99.4]
  Rubella: number analyzed (Participants) | 352 | 199
  Rubella | 86.4 [82.3 to 89.8] | 83.9 [78.1 to 88.7]
  VZV gE | 97.3 [95.0 to 98.7] | 97.5 [94.3 to 99.2]

ADVERSE EVENTS:
Time Frame: Solicited AEs: Day 1 to Day 7 post each vaccination, Solicited systemic AEs of salivary gland swelling, fever and rash: Day 1 to Day 30 post fourth vaccination; Unsolicited AEs: Day 1 to Day 30 post each vaccination. All-cause mortality, SAEs, AEs leading to withdrawal, AESIs and MAAEs: For participants not reaching Day 481 by Protocol Amendment 7: first vaccination (Day 1) to Day 481, for participants past Day 481 by the amendment: first vaccination (Day 1) to Day 661
Arm/Group | MenB+PCV Group | Placebo+PCV Group
All-Cause Mortality (participants affected / at risk) | 0/781 | 0/403
Serious Adverse Events (participants affected / at risk) | 35/781 | 19/403
Other Adverse Events (participants affected / at risk) | 771/781 | 389/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenB+PCV Group (N=781) | Placebo+PCV Group (N=403)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bronchogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
PFAPA syndrome (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 4 (4) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Picornavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 (3) | 2 (2)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 3 (3) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenB+PCV Group (N=781) | Placebo+PCV Group (N=403)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 20 (21) | 20 (23)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Brachycephaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Craniofacial deformity (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Kidney duplex (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Macrocephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Plagiocephaly (Congenital, familial and genetic disorders) | 3 (3) | 3 (3)
Strabismus congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Tethered oral tissue (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Conductive deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 9 (9) | 5 (5)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Astigmatism (Eye disorders) | 1 (1) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 3 (3) | 1 (1)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 3 (3)
Eye movement disorder (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 2 (2) | 1 (2)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Eyelid rash (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Pseudostrabismus (Eye disorders) | 1 (1) | 0 (0)
Scleral discolouration (Eye disorders) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 31 (32) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 334 (350) | 178 (193)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (4) | 1 (1)
Food protein-induced enterocolitis syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 (14) | 9 (9)
Gastrooesophageal reflux in neonate (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Infantile spitting up (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 75 (84) | 46 (55)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 317 (328) | 159 (174)
Vomiting projectile (Gastrointestinal disorders) | 1 (1) | 1 (1)
Administration site erythema (General disorders) | 460 (460) | 170 (170)
Administration site induration (General disorders) | 480 (480) | 180 (180)
Administration site pain (General disorders) | 582 (582) | 201 (201)
Administration site swelling (General disorders) | 322 (322) | 122 (122)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Adverse food reaction (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1)
Crying (General disorders) | 432 (433) | 163 (163)
Fatigue (General disorders) | 2 (2) | 2 (2)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Induration (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 0 (0)
Injection site bruising (General disorders) | 6 (6) | 6 (6)
Injection site discolouration (General disorders) | 1 (1) | 0 (0)
Injection site dryness (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0)
Injection site laceration (General disorders) | 0 (0) | 1 (1)
Injection site nodule (General disorders) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 2 (2) | 2 (6)
Injection site reaction (General disorders) | 1 (2) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Injection site urticaria (General disorders) | 1 (2) | 0 (0)
Injury associated with device (General disorders) | 1 (1) | 0 (0)
Irritability postvaccinal (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 521 (543) | 172 (184)
Swelling (General disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1)
Tenderness (General disorders) | 1 (1) | 0 (0)
Vaccination site bruising (General disorders) | 0 (0) | 1 (1)
Vaccination site irritation (General disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 5 (5) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 2 (3) | 1 (2)
Body tinea (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 30 (31) | 13 (16)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Bullous impetigo (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 6 (6) | 5 (5)
Candida infection (Infections and infestations) | 5 (5) | 0 (0)
Candida nappy rash (Infections and infestations) | 10 (11) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 17 (20) | 15 (17)
Conjunctivitis bacterial (Infections and infestations) | 4 (4) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1)
Coxsackie viral infection (Infections and infestations) | 2 (2) | 1 (1)
Croup infectious (Infections and infestations) | 24 (25) | 3 (4)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 4 (4) | 0 (0)
Erythema infectiosum (Infections and infestations) | 2 (2) | 0 (0)
Exanthema subitum (Infections and infestations) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (2)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 8 (8) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 9 (9) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 7 (7) | 3 (3)
Impetigo (Infections and infestations) | 3 (4) | 3 (3)
Influenza (Infections and infestations) | 13 (13) | 3 (3)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngotracheitis obstructive (Infections and infestations) | 2 (2) | 2 (2)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 40 (46) | 18 (20)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 5 (5) | 4 (4)
Oral viral infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 47 (55) | 29 (37)
Otitis media acute (Infections and infestations) | 33 (42) | 23 (28)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1)
Parvovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pustule (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 (3) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 9 (9) | 3 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 5 (5) | 0 (0)
Roseola (Infections and infestations) | 2 (2) | 1 (1)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 6 (6)
Skin candida (Infections and infestations) | 5 (5) | 3 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 125 (149) | 62 (79)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Viral infection (Infections and infestations) | 13 (14) | 7 (7)
Viral pharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Viral rash (Infections and infestations) | 3 (3) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 16 (17) | 12 (12)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Accident at home (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scrotal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood lead increased (Investigations) | 0 (0) | 1 (1)
Body temperature decreased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 2 (2) | 2 (2)
Human rhinovirus test positive (Investigations) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 2 (2)
Serum ferritin decreased (Investigations) | 1 (1) | 4 (4)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Breast milk substitute intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 543 (544) | 216 (217)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Milk soy protein intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Jaw clicking (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Drooling (Nervous system disorders) | 0 (0) | 1 (1)
Fine motor delay (Nervous system disorders) | 1 (1) | 0 (0)
Infant irritability (Nervous system disorders) | 2 (2) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Movement disorder (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 681 (681) | 319 (322)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 1 (1)
Breath holding (Psychiatric disorders) | 1 (1) | 0 (0)
Dependent personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5)
Irritability (Psychiatric disorders) | 713 (738) | 330 (345)
Middle insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Selective eating disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Renal hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Single functional kidney (Renal and urinary disorders) | 1 (1) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital labial adhesions (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Penile cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile dermatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Brief resolved unexplained event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 51 (58) | 20 (25)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 39 (44) | 17 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (5)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 31 (39) | 17 (20)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 25 (27) | 12 (14)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acne infantile (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 38 (41) | 22 (25)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 16 (16) | 10 (10)
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 216 (224) | 106 (117)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (4)
Child abuse (Social circumstances) | 1 (1) | 0 (0)
Cyanosis (Vascular disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 3 (3) | 1 (1)
Scalp haematoma (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT03621670/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT03621670/SAP_001.pdf